CLINICAL TRIAL: NCT07075445
Title: Observational Study to Describe Health-Related Quality of Life and Disease Burden Among Patients With Long QT Syndrome (LQTS) 2 and 3
Brief Title: Observational Study to Describe Health-Related Quality of Life and Measure Disease Burden Among Patients With Long QT Syndrome Types (LQTS) 2 and 3
Status: Recruiting | Type: Observational
Sponsor: Thryv Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Thryv Therapeutics Inc.
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Long QT Syndrome Type 3; Long QT Syndrome 2
MeSH Terms: conditions — Long QT syndrome type 3; Long Qt Syndrome 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional observational study designed to assess the disease burden and quality of life in individuals with LQTS 2 and 3. Each participant will answer each patient-reported outcome questionnaire only once over a 6-month period. The study will enroll up to 200 participants.

DETAILED DESCRIPTION:
The aim of the present cross-sectional observational study is to evaluate the health status and quality of life burden in patients with LQTS. The total study duration is anticipated to last for a period of up to 18 months, including up to 6 months of each individual's observation period. The observation period may be extended by up to 3 months (total 9 months). During the optional extension, data collection via myQTwave will be limited to emotional and physical symptoms survey. This prospective cohort study will collect PRO information in a cohort of patients with LQTS 2 or 3. All screened participants will be assigned a unique identifier. Eligible participants will download the myQTwave app on the Apple iPhone and Apple Watch delivered to them after enrollment.

Patient-reported outcomes will be captured via the Apple iPhone and daily health metrics (sleep, physical and Heart-related data) will be collected using the Apple Watch.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is willing and provides written informed consent to participate in this study.
2. Male or female participant of at least 18 years of age, English-speaking.
3. Confirmed genetic diagnosis of LQT2 or 3, demonstrated by one of the following:

   * Genetic testing report (pathogenic or likely pathogenic (P/LP) mutation) in KCHN2 or SCN5a genes) or,
   * A signed physician's letter confirming genetic diagnosis of LQTS 2 or 3.
4. Documented QTc ≥ 480 ms within the last year, demonstrated by one of the following:

   * 12-lead electrocardiogram (ECG), or
   * A signed physician's letter confirming an ECG demonstrating QTc value ≥ 480 ms.
5. The participant is able to operate a smartphone and a companion watch. *The number of participants with QTc between 480 and 500 ms will be limited to 50.

Exclusion Criteria:

1. Current participation in another clinical trial involving a drug or device.
2. Participants unwilling to use an iPhone or Apple Watch for the duration of the study.
3. Known diagnosis of Brugada Syndrome
4. Participants unwilling to comply with outlined procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from cardiology and genetic clinics at academic and private medical centers across the United States, as well as through outreach efforts targeting individuals and families affected by inherited arrhythmia conditions. This includes engagement through community-based initiatives. The study population includes individuals with a genetically confirmed diagnosis of Long QT Syndrome type 2 or 3.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) | Month 1
  Score from the Satisfaction With Life Scale (SWLS)
Quality of Life (QoL) | Month 1
  Score from the Quality of Life in Life-Threatening Illness - Late Adolescents and Adults Scale (QOL-LAS)
Disease burden | Month 2
  Score from the CDC HRQOL-4 (Health-Related Quality of Life)
Disease burden | month 2
  Score from the self-reported NYHA (New York Heart Association Classification)
Disease burden | Month 2
  Score from the Health Actions Evaluation (HAE-10)
Illness perception | Month 3
  Score from the Brief Illness Perception Questionnaire (B-IPQ)
Illness perception | Month 3
  Score from the Illness Intrusiveness Questionnaire (IIQ)
Psychosocial health, including distress, social and psychological well-being, and cardiac-specific measures, | Month 4
  Score from the Depression, Anxiety, and Stress Scale-21 (DASS-21)
Psychosocial health, including distress, social and psychological well-being, and cardiac-specific measures, | Month 4
  Score from the UCLA 3-Item Loneliness Scale
Psychosocial health, including distress, social and psychological well-being, and cardiac-specific measures, | Month 3
  Score from the Multidimensional Scale of Perceived Social Support (MSPSS)

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Greenville, North Carolina, United States